CLINICAL TRIAL: NCT06037876
Title: Efficacy of the Combination Ivermectin and Albendazole vs Albendazole Alone in School-aged Children Infected With Trichuris Trichiura: a Randomized Controlled Trial
Brief Title: Efficacy of Ivermectin-albendazole vs Albendazole Alone in School-aged Children Infected With Trichuris Trichiura
Acronym: FACEITeffic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Vector Borne & Neglected Tropical Disease Control Division, Ministry of Health, Uganda (Unknown)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRCCH PII 2021
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Trichuriasis
Keywords: Soil-transmitted helminths, Trichuris trichiura
MeSH Terms: conditions — Trichuriasis | interventions — Intravital Microscopy; Albumins; Albendazole; Ivermectin

STUDY DESIGN:
Intervention Model Description: Parallel open-label randomized controlled superiority trial
Who Masked: Outcomes Assessor
Masking Description: Allocation concealment will be warranted using sequential, opaque, sealed envelopes. Outcome assessors in the lab will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVM (200 µg/kg) + ALB (400 mg) (Experimental): A single tablet of albendazole (400mg) plus 200 µg/kg of ivermectin, provided as single oral dose.
  Interventions: Drug: IVM (200 µg/kg) + ALB (400 mg)
- ALB (400mg) (Active Comparator): A single tablet of albendazole (400mg), provided as single oral dose.
  Interventions: Drug: ALB (400mg)

INTERVENTIONS:
Drug: IVM (200 µg/kg) + ALB (400 mg) — World Health Organization Pre-Qualification (WHO PQ) recommended ivermectin 3mg tablets will be used together with albendazole 400mg tablets as provided by WHO for Neglected Tropical Disease (NTD) programs.
  Other Names: Zentel® and Stromectol®, Ivermectin Tablet 3mg
  Arms: IVM (200 µg/kg) + ALB (400 mg)
Drug: ALB (400mg) — Albendazole 400mg manufactured and donated by GlaxoSmithKline (GSK) to WHO
  Other Names: Zentel®
  Arms: ALB (400mg)

SUMMARY:
The goal of this parallel open-label randomized controlled superiority trial is to demonstrate that co-administered ivermectin (200 µg/kg) plus albendazole (400 mg) is superior to albendazole (400 mg) monotherapy in terms of cure rates against Trichuris trichiura infections assessed by Kato-Katz at 14-21 days post-treatment in individuals aged 6-12 years.

The main questions it aims to answer are:

* Is single oral dose combined ivermectin-albendazole superior to albendazole alone in terms of cure rates and egg reduction rates against T. trichiura infections in children aged 6-12 years in Uganda?
* Is single oral dose combined ivermectin-albendazole superior to albendazole alone in terms of cure rates and egg reduction rates against co-infecting soil-transmitted helminth infections such as Ascaris lumbricoides and hookworm in children aged 6-12 years in Uganda?
* Is single oral dose combined ivermectin-albendazole as tolerable and safe as albendazole monotherapy in children aged 6-12 years in Uganda?

Participants will be asked to provide two stool samples at baseline that will be subjected to microscopic analysis using the Kato-Katz thick smear technique for detection of soil-transmitted helminth eggs. T. trichiura-infected participants will be:

* clinically examined for general health, anthropometric parameters including height and weight as well as temperature
* randomly assigned to either receive one single oral dose of combined ivermectin and albendazole or albendazole monotherapy
* checked for any potential adverse events and will undergo a brief questionnaire on specific symptoms 3h after drug administration
* asked to provide another two stool samples to be microscopically examined for helminth eggs 14-21 days post-treatment Researchers will compare individuals treated with ivermectin-albendazole and albendazole alone to see if the proportion of T. trichiura egg-negative individuals and/or reduction in egg counts differs between these two groups 14-21 days after treatment.

DETAILED DESCRIPTION:
In view that efficacy of co-administered ivermectin (IVM) and albendazole (ALB) has been found to vary between different settings the rationale of this parallel open-label randomized controlled superiority trial is to provide evidence on the efficacy of co-administered ivermectin and albendazole compared to albendazole monotherapy in school-aged children aged 6-12 years against infection with T. trichiura in Uganda.

Our primary objective is to demonstrate superiority of

1. Arm A: single dose of ivermectin (200 µg/kg, 3 mg tablets according to weight) / single dose of albendazole (400 mg tablet) combination, compared to
2. Arm B: single dose of albendazole (400 mg tablet)

in terms of cure rate (CR) against T. trichiura infections in school-aged children aged 6-12 years assessed at 14-21 days post-treatment by Kato-Katz microscopy.

The secondary objectives of the trial are:

1. to determine the egg reduction rates (ERRs) of ivermectin/albendazole combination therapy compared to albendazole monotherapy against T. trichiura
2. to determine the CRs and ERRs of the study drugs against Ascaris lumbricoides and hookworm in co-infected participants
3. to evaluate the safety and tolerability of the treatment

The study will be implemented as a school-based study and children aged 6-12 years from two primary schools in Kabale district, southwestern Uganda will be invited for parasitological examination after obtaining informed consent from parents/caregivers and assent by the minor participants. Two stool samples will be collected, when possible, on two consecutive days. Children found to be infected with T. trichiura based on quadruplicate Kato-Katz thick smear readings will be enrolled into the actual trial. The medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study nurse/physician before treatment.

All participants will be interviewed before treatment and after 3 and 24 hours (active surveillance) for the occurrence of adverse events (AEs). Participants and their caregivers will be told that any potential AEs happening between 24 hours and the respective follow-up time point for stool collection should be reported to the local village health team (VHT) members, which will be trained to handle the situation by taking the participant to a health facility for timely treatment, or to local health workers directly.

The efficacy of the treatment will be determined at 14-21 days post-treatment by collecting another two stool samples.

At both, baseline and follow-up (14-21 days post treatment) a portion of stool (1.5-2 g) from all participants identified with T. trichiura infections will be preserved in 95% ethanol, shipped to a reference laboratory in Switzerland and subjected to amplicon deep sequencing for characterization of T. trichiura strains and investigation of potential resistance markers.

Study participants eligible for treatment will be randomly assigned to one of the two treatment arms stratified by 2 levels of baseline infection intensity (light: 1-999 EPG, and moderate plus heavy: ≥ 1000 EPG T. trichiura infections).

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, a per-protocol analysis will be conducted. CRs will be calculated as the percentage of egg-positive subjects at baseline who become egg-negative after treatment. Differences among CRs (between treatment arms) will be analyzed by using crude and adjusted logistic regression modeling.

Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for differences in ERRs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation signed from caregivers; and written assent by participants.
* Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and at follow-up assessment 14-21 days after treatment.
* Willing to be examined by a study nurse/physician prior to treatment.
* At least two slides of the quadruple Kato-Katz thick smears positive for T. trichiura.

Exclusion Criteria:

* Presence or signs of major systemic illnesses, e.g. body temperature ≥ 38°C, clinical malaria (fever + positive RDT) upon initial clinical assessment.
* Recent use of anthelmintic drug (within past 4 weeks).
* Attending other experimental research studies.
* Known allergy to study medications (i.e. benzimidazole or ivermectin).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants T. Trichiura Egg Negative Post-Treatment (Cured) | 14-21 days after treatment
  The conversion from being egg positive pre-treatment to egg negative post-treatment, or cure rate (CR).

SECONDARY OUTCOMES:
Egg Reduction Rate (ERR) against T. Trichiura | 14-21 days after treatment
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Number of Participants With Concomitant Soil-transmitted Helminth Infections Egg Negative Post-Treatment (Cured) | 14-21 days after treatment
  Number of participants that converted from egg positive with Ascaris lumbricoides and/or hookworm infections to egg negative after 14-21 days.
Egg-reduction Rates (ERRs) Against Concomitant Soil-transmitted Helminth Infections | 14-21 days after treatment
  Percent change in geometric mean eggs per gram of stool from before to after treatment. ERRs will be calculated for Ascaris lumbricoides and hookworm infections as described in outcome 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Vector Borne & Neglected Tropical Disease Control Division, Ministry of Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmeirim MS, Hurlimann E, Beinamaryo P, Kyarisiima H, Nabatte B, Hattendorf J, Steinmann P, Keiser J. Efficacy and safety of albendazole alone versus albendazole in combination with ivermectin for the treatment of Trichuris trichiura infections: An open-label, randomized controlled superiority trial in south-western Uganda. PLoS Negl Trop Dis. 2024 Nov 26;18(11):e0012687. doi: 10.1371/journal.pntd.0012687. eCollection 2024 Nov. PMID 39591454